CLINICAL TRIAL: NCT05608265
Title: Scanning Laser Ophthalmoscopy Registered Optical Coherence Tomography for Real-Time Eye Tracking
Brief Title: Real-time Eye Tracking and Imaging of the Eye in Diabetic Retinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseMedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OSNATFIHIO001
Record Dates: First submitted 2022-09-26; First posted 2022-11-08 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Retinopathy; Retinal Imaging
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinal Imaging using the OSNAT800 IO device (Experimental): Patients will have their eyes imaged with the OSNAT800 IO device in addition to a routine standard of care appointment.
  Interventions: Device: OSNAT 800 IO

INTERVENTIONS:
Device: OSNAT 800 IO — Real-time, combined scanning laser ophthalmoscope (SLO) and optical coherence tomography (OCT) for retinal imaging

SUMMARY:
Diabetic retinopathy (DR) is a leading cause of vision loss in working age Canadians. Current treatment consists of early detection and laser photocoagulation therapy for preventing progressive or severe vision loss. Microaneurysms (MA) are the earliest, clinically visible changes of DR, which are visualized using specialized imaging technologies. PulseMedica is developing a three-dimensional (3D) retinal imaging system with real-time eye tracking capabilities. The purpose of this study is to assess the feasibility of PulseMedica's prototype device, the OSNAT800 Imaging Only (IO), in providing real-time tracking of eye movements in patients with DR. It is hypothesized that the OSNAT 800 IO will be able to perform real-time eye tracking while imaging patients with DR.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years of age
* Male or female
* Diagnosed diabetic retinopathy
* Two eyes with clear ocular media

Exclusion Criteria:

* Patients younger than 18 years and over 70 years of age
* Patients without diabetic retinopathy
* Opacification of cornea, lens, or vitreous

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Successful performance of the real-time eye tracking function by post-image processing | Through study completion, an average of 6 months
  Successful acquisition of retinal images

SECONDARY OUTCOMES:
Device usability as assessed by a survey | Through study completion, an average of 6 months
  Qualitative assessment of user feedback
Image Quality as assessed by user assessment of image quality parameters | Through study completion, an average of 6 months
  Qualitative assessment of image at time of acquisition

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Retina Consultants, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No